CLINICAL TRIAL: NCT00676923
Title: LABS-3 Diabetes: Mechanisms for Improvement of Type 2 Diabetes Following Bariatric Surgery
Brief Title: Improving Diabetes After Bariatric Surgery
Acronym: LABS-3
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: DK6657_3b; U01DK066557 (NIH)
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this project is to examine the physical mechanisms that contribute to improvements of glucose tolerance in type 2 diabetes mellitus (DM) following certain types of bariatric surgery.

DETAILED DESCRIPTION:
The goal of this project is to examine the physiological mechanisms that contribute to improvements of glucose homeostasis in type 2 diabetes mellitus (DM) following gastric bypass Roux-en-Y bariatric surgery (GBP). The central hypotheses are: 1) that surgical changes in the anatomy of nutrient absorption achieved by GBP change incretin hormone secretion which in turn improves pancreatic islet function; and 2) that improvement in insulin secretion induced by the changes in incretin function, together with improvement in insulin resistance induced by weight loss, normalize glucose homeostasis in type 2 DM.

Funds are not available to pay for the surgery for patients, only to address research questions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age and undergo bariatric surgery by a LABS certified surgeon.
* Enrollment in LABS-1 or LABS-2.
* Documented type 2 diabetes (fasting plasma glucose greater than 125 mg/dl) that is treated with lifestyle efforts (drug naïve) or taking acceptable oral medications (see appendix) with a HgA1c less than or equal to 8.5% and a fasting blood glucose less than or equal to 180 mg/dL. This will be one group.
* Non-diabetic (ND) with normal values for fasting glucose and HbA1c. This will be the second group.
* Adequate IV access.

Exclusion Criteria:

* Informed consent not obtained.
* Patient with diabetes with an HbA1c greater than 8.5% or a fasting blood glucose greater than 180 mg/dL.
* Creatinine greater than 1.7.
* Unlikely to comply with the 6 month follow-up (post-surgical) protocol (i.e. geographically inaccessible for study visits) or unable to communicate with local study staff.
* Use of unacceptable diabetic medications (see appendix) at baseline (see appendix).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from the LABS-2 cohort at participating LABS clinical centers.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2008-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Purnell, MD, Study Director — Oregon Health and Science University
Locations (5):
- United States (5):
  - Legacy Good Samaritan Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- See also: Related Info — http://www.niddklabs.org